CLINICAL TRIAL: NCT02826772
Title: A Phase 1/2, Multi-Center, Open-Label, Two-Stage Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of GT0918 in Subjects With Metastatic Castrate Resistant Prostate Cancer (mCRPC)
Brief Title: Safety, Tolerability, and PK of GT0918 (Proxalutamide) in Subjects With Metastatic Castrate Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Kintor Pharmaceutical Inc, (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GT0918-US-1001
Record Dates: First submitted 2016-06-23; First posted 2016-07-11 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Metastatic Castrate Resistant Prostate Cancer (mCRPC)
MeSH Terms: interventions — proxalutamide; Androgen Receptor Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phase 1 GT0918 level 1 (Experimental): generic name: not applicable dosage form: tablet dosage: oral dosage to be determined dosage frequency: daily dosage duration: 6 months
  Interventions: Drug: GT0918

INTERVENTIONS:
Drug: GT0918 — anti-tumor activity
  Other Names: androgen receptor antagonist; proxalutamide

SUMMARY:
This was a Phase 1, multicenter, open-label, clinical trial in adult subjects with metastatic castrate resistant prostate cancer who progressed after both hormonal therapy (abiraterone or enzalutamide) and chemotherapy (docetaxel), or cannot tolerate either or both therapies.

The study involved a Phase 1 dose escalation of oral GT0918 to evaluate its safety, tolerability, pharmacokinetics and pharmacodynamics.

DETAILED DESCRIPTION:
GT0918 treatment was initiated with the first dose of 50 mg/day in a cohort of 3 patients, and 6- patients per cohort for the subsequent escalated dose levels at 100 mg, 200 mg, 300 mg, 400 mg, 500 mg and 600 mg/day. Patients received orally administered GT0918 once daily at the indicated doses for 28 consecutive days (4 weeks), followed by a 7-day off-treatment period for PK analysis. This concluded the Cycle 1 treatment. Patients who could not complete the first cycle of 28 days for DLT evaluation were to be considered as early termination and replaced. Upon completion of the Cycle 1 treatment, if no DLT occurred in the cohort of 3 patients, or no more than 1 patient had DLT in cohorts with at least 6 patients, dose escalation was allowed for the subsequent higher dose.

Patients were to receive up to 6 cycles of GT0918 treatments at their assigned dose levels if they were evaluated by the investigator to have no unacceptable toxicity and show evidence of clinical benefit (stable disease or a response) per RECIST v1.1 criteria and PSA assessments. No off-treatment periods were scheduled for the additional cycles from Cycle 2 beyond. Patients had to be evaluated bi-monthly for their eligibility to continue the treatment of additional cycles. Patient evaluations included CT and/or MRI scans performed every 2 cycles (8 weeks), as well as physical examinations, ECOG performance status, PSA measurements, which were performed every 4 weeks. Cycles beyond the 6th cycle were optional for eligible subjects that did not exhibit progressive disease (PD). Eligible patients could be treated for a total of 6 months at their assigned dose level at the investigator's discretion.

Patients would have an End-of-Study (EOS) visit if treatment were discontinued due to intolerable toxicities, disease progression, withdrawal of consent. Safety follow-up for possible delayed drug-related AE or side effects can be performed by phone call or office visit if needed.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to any study-related procedure being performed.
2. Subjects at least 18 years of age or older at the time of consent.
3. Histologically confirmed metastatic castrate resistant cancer (mCRPC) who progressed after both hormonal therapy (abiraterone or enzalutamide) and chemotherapy (docetaxel, for example); or cannot tolerate either or both of these classes of therapies.
4. Ongoing androgen deprivation therapy with a luteinizing hormone-releasing hormone (LHRH) "super-agonist" or antagonist, or bilateral orchiectomy and serum testosterone level < 50 ng/dL (< 0.5 ng/mL, < 1.7 nmol/L) at screening.
5. Metastatic disease documented by computed tomography (CT)/magnetic resonance imaging (MRI) or bone scan.
6. Progressive disease despite ongoing androgen deprivation or chemotherapy. Progressive disease is defined by 1 or more of the following criteria:

   * Subjects with a rising PSA value > 2 ng/mL in at least 2 measurements, at least 1 week apart. If the confirmatory PSA value is less than the screening PSA value, then an additional test for the rising PSA is required to document progression.
   * Subjects with measurable disease, progression defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.
   * Subjects with metastatic bone disease, progression defined by 2 or more new lesions in a radionuclide bone scan.
7. ECOG performance status of 0-2 (dose escalation phase); ECOG performance status of 0-1 (expansion phase).
8. Screening blood counts of the following:

   * Absolute neutrophil count ≥ 1500/μL
   * Platelets ≥ 100,000/μL
   * Hemoglobin > 9 g/dL
9. Screening chemistry values of the following:

   * Alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤ 2.5 × upper limit of the normal reference range (ULN)
   * Total bilirubin ≤ 2 × ULN
   * Creatinine ≤ 1.5 × ULN
   * Albumin > 2.8 g/dL.
10. At screening, life expectancy of at least 3 months.
11. Subjects whose partners are women of childbearing potential (WOCBP) must use an adequate method of birth control while on study drug and at least for 3 weeks after discontinuation of study drug.
12. Subject is willing and able to comply with all protocol required visits and assessments.

Exclusion Criteria:

1. Subjects with life expectancy less than 3 months.
2. Discontinuation of bicalutamide or nilutamide less than 6 weeks, and other antiandrogens less than 4 weeks, abiraterone less than 3 weeks, prior to the start of study medication.
3. Prior chemotherapy, radiation, sipuleucel-T or other experimental immunotherapy less than 4 weeks prior to the start of study medication.
4. Prior chemotherapies more than 2 lines (Phase II part only) .
5. Ongoing acute treatment-related toxicity associated with a previous therapy greater than grade 1 except for grade 2 alopecia or neuropathy.
6. History of impaired adrenal gland function (eg, Addison's disease, Cushing's syndrome).
7. Known gastrointestinal disease or condition that affects the absorption of GT0918.
8. History of congestive heart failure New York Heart Association (NYHA) class III or IV or uncontrolled hypertension at screening.
9. History or family history of long QT syndrome.
10. History of other malignancy within the previous 3 years, except basal cell or squamous cell carcinoma, or non-muscle invasive bladder cancer.
11. Use of systemic glucocorticoid (eg, prednisone, dexamethasone) within 14 days prior to the start of study medication.
12. Co-administration of CYP3A4 ligands that serve as substrates or induce or inhibit the enzyme.
13. Prior use of any herbal products known to decrease PSA levels (eg, PC-SPES or saw palmetto) within 30 days prior to the start of study medication.
14. Major surgery within 30 days prior to the start of study medication.
15. Blood transfusion (including blood products) within 1 week of screening.
16. Serious persistent infection within 14 days prior to the start of study medication.
17. Serious concurrent medical condition including CNS disorders.
18. Previous history of difficulty swallowing capsules.
19. Known hypersensitivity to GT0918 or its excipients.
20. Any condition that, in the opinion of the investigator, would impair the subject's ability to comply with study procedures.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-02-10 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
dose-limiting toxicities (DLTs) | 1 month
  abnormal laboratory value
maximum tolerated dose (MTD),biological dose or minimal effective dose, (MED), and recommended Phase 2 dose(s) (RP2D). | 1 month
  50 mg, 100 mg, 200 mg, 300 mg, 400 mg or 500 mg of GT0918

SECONDARY OUTCOMES:
maximum concentration (Cmax) | 6 months
  Pharmacokinetics
time that maximum concentration is observed (tmax) | 6 months
  Pharmacokinetics
area under the concentration time-curve from time zero to infinity (AUC0∞) | 6 months
  Pharmacokinetics
area under the plasma concentration-time curve from time zero hours to time (t hrs), (AUC0-t) | 6 months
  Pharmacokinetics
area under the plasma concentration-time curve from time zero hours to 24 hours (AUC0-24) | 6 months
  Pharmacokinetics
terminal elimination rate constant (λz) | 6 months
  Pharmacokinetics
terminal elimination half life (t½) | 6 months
  Pharmacokinetics
volume of distribution (Vz) | 6 months
  Pharmacokinetics
volume of plasma cleared of the drug per unit time (C) | 6 months
  Pharmacokinetics
circulating tumor deoxyribonucleic acid (ctDNA) | 6 months
  antitumor activities
circulating messenger ribonucleic acid (mRNA) | 6 months
  antitumor activities
circulating tumor cells (CTC) | 6 months
  antitumor activities
prostate-specific antigen (PSA) | 6 months
  biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Phoebe Zhang, PhD, Study Director — Suzhou Kintor Pharmaceuticals, Inc.
Locations (6):
- United States (6):
  - Chesapeake Urology Research Associates, Towson, Maryland
  - G U Research Network, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Rutgers University, New Brunswick, New Jersey
  - North Shore Hematology Oncology Associates, East Setauket, New York
  - Gabrail Cancer Center Research, Canton, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maia MC, Salgia M, Pal SK. Harnessing cell-free DNA: plasma circulating tumour DNA for liquid biopsy in genitourinary cancers. Nat Rev Urol. 2020 May;17(5):271-291. doi: 10.1038/s41585-020-0297-9. Epub 2020 Mar 17. PMID 32203306